CLINICAL TRIAL: NCT01103310
Title: Open-label, Multi Center Study for an Evaluation of Radiation Dosimetry, Plasma Pharmacokinetics, Safety and Tolerability of the 18F-labeled PET/CT (Positron Emission Tomography / Computed Tomography) Tracer BAY94-9392 Following a Single Intravenous Administration of 300 MBq (Corresponding to ≤ 100 µg Total Quantity) in Healthy Volunteers, as Well as the Investigation of Safety, Tolerability, Pharmacokinetics, and Diagnostic Performance of the Tracer in PET/CT in Cancer Patients or Patients With Inflammation.
Brief Title: Radiation Dosimetry, Metabolism, Pharmacokinetics, Safety and Tolerability and PET Imaging With BAY94-9392 in Healthy Volunteers and Patients With Cancer or Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14207
Record Dates: First submitted 2010-03-31; First posted 2010-04-14 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Diagnostic Imaging; Neoplasms
Keywords: Neoplasm; PET/CT diagnosis; PET tracer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Cancer patients, single intravenous bolus injection of 300 MBq BAY94-9392 on day one of the treatment period, PET/CT
  Interventions: Drug: BAY94-9392
- Arm 2 (Experimental): Healthy volunteers, single intravenous bolus injection of 300 MBq BAY94-9392 on day one of the treatment period, whole body PET/CT for determination of effective dose, kinetics of BAY94-9392 in blood
  Interventions: Drug: BAY94-9392

INTERVENTIONS:
Drug: BAY94-9392

SUMMARY:
Visual assessment of diagnostic PET/CT (positron emission tomography/computed tomography) images obtained after a single intravenous injection of BAY94-9392 in patients with cancer or inflammation.

ELIGIBILITY:
Inclusion criteria:

In Germany Healthy volunteers

* Males/females ≥ 50 and ≤ 65 years Patients
* Males/females ≥ 35 and ≤ 75 years
* histologically confirmed diagnosis of non small cell lung cancer or adenocarcinoma of the breast with a positive FDG-PET or
* patient with primary prostate cancer scheduled for prostatectomy and patient with prostate tumor recurrence with a positive choline-PET, the initial disease is histologically confirmed or
* inflammation with a positive FDG-PET

In Korea Patients

* Males/females ≥ 35 and ≤ 75 years
* histologically confirmed diagnosis of non small cell lung cancer, adenocarcinoma of the breast or hepatocellular cancer with a positive FDG-PET or
* patient with primary prostate cancer scheduled for prostatectomy and patient with prostate tumor recurrence with a positive choline-PET, the initial disease is histologically confirmed or
* inflammation (positive FDG-PET mandatory, could be also done as screening examination)

Exclusion criteria:

* Concurrent severe and/or uncontrolled and/or unstable medical disease other than cancer or inflammation (e.g. poorly controlled diabetes, congestive heart failure, myocardial infarction within 12 months prior to planned injection of BAY 94-9392, unstable and uncontrolled hypertension, chronic renal or hepatic disease, severe pulmonary disease) which could compromise participation in the study
* Known sensitivity to the study drug or components of the preparation

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Visual assessment of lesion | Day of study drug administration

SECONDARY OUTCOMES:
Quantitative analysis of BAY94-9392 uptake into lesions (Standardized Uptake Values = SUVs) | Day of study drug administration
Electrocardiogram (ECG) | At least twice within 2 days after treatment
Blood pressure | At least twice within 2 days after treatment
Serum protein | At least twice within 2 days after treatment
Serum creatinine | At least twice within 2 days after treatment
Serum GOT (Glutamate-Oxalacetate-Transaminase) | At least twice within 2 days after treatment
Adverse events collection | Continuously for at least 4 days after treatment
Radiation doses per organ (µGy/MBq) | Day of study drug administration
Higher organ dose (HT) | Day of study drug administration
Doses per organ (µSv/MBq) | Day of study drug administration
Effective dose (µSv/MBq) | Day of study drug administration
Effective dose resulting from the total administered diagnostic activity of 300 MBq +/- 10% | Day of study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Stanford, California, United States
- München, Bavaria, Germany
- Seoul, South Korea

REFERENCES:
- [Background] Baek S, Mueller A, Lim YS, Lee HC, Lee YJ, Gong G, Kim JS, Ryu JS, Oh SJ, Lee SJ, Bacher-Stier C, Fels L, Koglin N, Schatz CA, Dinkelborg LM, Moon DH. (4S)-4-(3-18F-fluoropropyl)-L-glutamate for imaging of xC transporter activity in hepatocellular carcinoma using PET: preclinical and exploratory clinical studies. J Nucl Med. 2013 Jan;54(1):117-23. doi: 10.2967/jnumed.112.108704. Epub 2012 Dec 11. PMID 23232273
- [Background] Baek S, Choi CM, Ahn SH, Lee JW, Gong G, Ryu JS, Oh SJ, Bacher-Stier C, Fels L, Koglin N, Hultsch C, Schatz CA, Dinkelborg LM, Mittra ES, Gambhir SS, Moon DH. Exploratory clinical trial of (4S)-4-(3-[18F]fluoropropyl)-L-glutamate for imaging xC- transporter using positron emission tomography in patients with non-small cell lung or breast cancer. Clin Cancer Res. 2012 Oct 1;18(19):5427-37. doi: 10.1158/1078-0432.CCR-12-0214. Epub 2012 Aug 14. PMID 22893629
- [Background] Smolarz K, Krause BJ, Graner FP, Wagner FM, Hultsch C, Bacher-Stier C, Sparks RB, Ramsay S, Fels LM, Dinkelborg LM, Schwaiger M. (S)-4-(3-18F-fluoropropyl)-L-glutamic acid: an 18F-labeled tumor-specific probe for PET/CT imaging--dosimetry. J Nucl Med. 2013 Jun;54(6):861-6. doi: 10.2967/jnumed.112.112581. Epub 2013 Apr 8. PMID 23568366
- [Derived] Park SY, Na SJ, Kumar M, Mosci C, Wardak M, Koglin N, Bullich S, Mueller A, Berndt M, Stephens AW, Cho YM, Ahn H, Chae SY, Kim HO, Moon DH, Gambhir SS, Mittra ES. Clinical Evaluation of (4S)-4-(3-[18F]Fluoropropyl)-L-glutamate (18F-FSPG) for PET/CT Imaging in Patients with Newly Diagnosed and Recurrent Prostate Cancer. Clin Cancer Res. 2020 Oct 15;26(20):5380-5387. doi: 10.1158/1078-0432.CCR-20-0644. Epub 2020 Jul 21. PMID 32694158